CLINICAL TRIAL: NCT02164227
Title: EFFECTIVE USE OF RESPIRATORY PATTERNS IN THE FIRST PERIOD OF LABOR IN CONTROL OF MATERNAL ANXIETY: A CLINICAL TRIAL
Brief Title: Effective Use of Respiratory Patterns in the First Period of Labor in Control of Maternal Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Alessandra da Boaviagem Freire, Master student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 025972/2013
Record Dates: First submitted 2014-05-21; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety
Keywords: anxiety; breathing exercise; labour
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- respiratory pattern (Experimental): Deep and slow inspiration is used in the initial and active stages, at which time the contractions vary from uncomfortable to strong, lumbosacral pain and cervical dilation may occur between 3 and 8 cm in this case the mother is driven to inspire slowly and the level of inspiratory reserve volume followed by slow exhalation to functional residual capacity; Sigh with post-expiratory pause that corresponds to a small spontaneous exhalation to relax occurs in tidal volume; Expiratory delay that corresponds to a prolonged propelled with the lips during the lull and expiration in the expiration time that corresponds to a slow inspiration followed by two or three puffs with the short lips will be used propelled.
  Interventions: Other: Respiratory pattern
- Control (No Intervention): Follows the service routine

INTERVENTIONS:
Other: Respiratory pattern
  Arms: respiratory pattern

SUMMARY:
The effectiveness of breathing exercise on anxiety in women during the first period of labor.

DETAILED DESCRIPTION:
The groups will be randomized into intervention groups, which will be held ventilatory patterns while the control group will receive routine care service. The measurements will be made during the admission, and every 2 hours until the final phase of dilation.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* First stage of labor

Exclusion Criteria:

* Multiple gestation;
* Eclampsia;
* Pregnancy with a dead fetus;
* Use of analgesia;
* Pregnant women with clinical instability;
* Psychiatric disorders;

Ages: 12 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-07 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 2 hours
  The anxiety of patients will be assessed using IDATE questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Maternidade Professor Bandeira Filho, Recife, Pernambuco, Brazil